CLINICAL TRIAL: NCT05690958
Title: Dutch Population's Intended Uptake and Views on the Organization of Esophageal Cancer Screening: a Nationwide Survey
Brief Title: Public's Intended Uptake and Views on Organization of Esophageal Cancer Screening
Acronym: ACCEPT-survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 111597
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-01

CONDITIONS: Barrett Esophagus; Barrett Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Filling in a survey

SUMMARY:
Rationale: Research on novel methods to screen for esophageal adenocarcinoma (EAC) has expanded. Insight into individuals' drivers and barriers to attend screening is essential to tailor a potential new screening policy to their preferences. Public preferences should also be considered on the organizational level to guarantee client-centered decision-making in the design of the screening process.

Objective: This study will examine Dutch individuals' intended uptake of EAC screening, including factors that predict uptake, and their views on its organization.

Study design: Cross-sectional population-based survey. Study population: Dutch individuals aged 45-75 years. The required sample size is 2088 and 8350 individuals will be invited based on an assumed participation rate of 25%.

Methods: Eligible individuals will be selected from the Dutch population registry (BRP) using simple random sampling. Invitations will be sent by postal mail with participants being directed to a digital survey.

Main study parameters/endpoints: The primary outcome of the study is the intended uptake of EAC screening (strong vs weak). Secondary study endpoints are the perceived need for consultation, perceived need for general education campaigns, acceptability of risk stratification scenarios, and acceptability of using health care resources for EAC screening.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will not directly benefit from participating in this study. Nonetheless, participating in this study is not associated with any healthcare risks and the burden for the subjects is very low. The survey has a low burdensome nature and will take approximately 15 to 20 minutes to complete. All data will be pseudonymized, refusal to fill out the survey or desire to withdraw from the study will not have any consequences for the invited subject.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 to 75 years

Exclusion Criteria:

* Previous diagnosis of EAC.
* Unable to provide informed consent.
* Unable to fill out the digital survey.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are included in the study. We provide a non-binairy answer option for gender.
Study Population: A sample will be drawn from the Dutch population registry, the 'Basisregistratie Personen' (BRP), using simple random sampling.
Sampling Method: Probability Sample
Enrollment: 2088 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Intended uptake of EAC screening | Baseline
  Participants will be informed about BE/EAC screening. Participants will also be informed about using upper endoscopy for this purpose and 1 out of 3 alternative hypothetical screening scenario's (transnasal endoscopy, ingestible cell-collection device, or breath analysis. Subsequently, participants will be asked if they intend to attend upper endoscopy and the alternative test if they were invited.

SECONDARY OUTCOMES:
Views on the organization of EAC screening | Baseline
  Various items that are based on qualitative focus group results on the topic

OTHER OUTCOMES:
Age | Baseline
Gender | Baseline
Education | Baseline
Current GERD symptoms | 7 days
  Reflux Disease Questionnaire (RDQ)
Marital status | Baseline
Ethnicity | Baseline
Previous upper endoscopy experience | Baseline
Personal history of cancer | Baseline
Knowing someone affected by esophageal cancer | Baseline
General cancer worry | Baseline
  Lerman's cancer worry scale (CWS)
Perceived risk of EAC | Baseline
  Item adapted from HINTS survey
General screening intent and beliefs about cancer screening | Baseline
  Item adapted from screening module of awareness and beliefs about cancer (ABC) measure
Anticipated discomfort during the screening test | Baseline
  7-point Likert scale
Acceptability of screening test accuracy | Baseline
  7-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sijben J, Rainey L, Maas F, Broeders MJM, Siersema PD, Peters Y. The Public's Intended Uptake of Hypothetical Esophageal Adenocarcinoma Screening Scenarios: A Nationwide Survey. Am J Gastroenterol. 2024 Sep 1;119(9):1802-1812. doi: 10.14309/ajg.0000000000002812. Epub 2024 Apr 15. PMID 38619114